CLINICAL TRIAL: NCT05988619
Title: Combined Internet-Based Cognitive Behavioral Therapy With Transcranial Magnetic Stimulation for Patients With Major Depressive Disorder
Brief Title: iCBT With TMS in Patients With MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ben Rosenberg, Postdoctoral Fellow, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19000581
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder
Keywords: Depression; TMS; Brain Stimulation; Internet-Based CBT
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Care providers administering the TMS treatment are blinded and do not know whether the participant has been randomized to receive iCBT or educational content as a supplement to the TMS treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- iCBT and TMS (Active Comparator): All participants complete six weeks of TMS treatment (five days per week) within the UCLA TMS Clinic. Participants in this condition additionally access iCBT materials and attend a weekly session for 30 minutes with a trained mental health coach to discuss iCBT content.
  Interventions: Device: Transcranial Magnetic Stimulation; Behavioral: Internet-Based Cognitive Behavioral Therapy
- Psychoeducation and TMS (Placebo Comparator): All participants complete six weeks of TMS treatment (five days per week) within the UCLA TMS Clinic. Participants in this condition additionally access educational materials about mental health and attend a weekly session for 30 minutes with a trained mental health coach to discuss educational content.
  Interventions: Device: Transcranial Magnetic Stimulation; Behavioral: Psychoeducation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — TMS is a noninvasive method of brain stimulation administered by physicians in the UCLA TMS Clinical and Research Service. It is an FDA-approved treatment for Major Depressive Disorder.
  Other Names: TMS
Behavioral: Internet-Based Cognitive Behavioral Therapy — This Way Up is an internet-based cognitive behavioral therapy (iCBT) for depression and anxiety. Participants learn about depression and anxiety symptoms, as well as behavioral strategies for addressing these symptoms. Participants are provided with homework exercises designed to help them engage in these strategies regularly.
  Other Names: iCBT; This Way Up
  Arms: iCBT and TMS
Behavioral: Psychoeducation — Stories of the Mind is an educational program that is freely available through the Public Broadcast Service (PBS). Participants view video testimonials in which individuals describe their personal experiences across a variety of mental health concerns.
  Other Names: Stories of the Mind
  Arms: Psychoeducation and TMS

SUMMARY:
Major Depressive Disorder (MDD) is a common mental health diagnosis. While there are many approaches to the treatment of MDD, current treatments of MDD often do not substantially reduce depressive symptoms among those in need of care. Prior research suggests that combining cognitive-behavioral therapy (CBT) and psychopharmacology can produce optimal treatment outcomes compared to the use of either treatment individually. Transcranial Magnetic Stimulation (TMS) is one promising brain stimulation approach used to treat MDD, especially among patients with treatment-resistant symptoms. Like psychopharmacological interventions, TMS may produce optimal treatment outcomes when paired with CBT. However, standard TMS protocols are time-intensive, typically requiring daily doctor visits for one hour of six to eight weeks. Therefore, an internet-delivered CBT protocol may augment the effects of TMS without substantially increasing patient burden. To that end, the present study assesses if a combined TMS and internet-delivered CBT protocol may produce superior treatment outcomes compared with TMS alone.

ELIGIBILITY:
Inclusion Criteria:

Subjects with Major Depressive Disorder who are receiving a full course of TMS treatment in at the UCLA TMS Clinic. Eligibility is determined by TMS physicians who are co-investigators on this study.

Exclusion Criteria:

Any indications of metal implants, pregnancy, psychosis, autism spectrum disorders, complex regional pain syndromes, substance use dependence and comorbidities that would interfere with treatment response. The criteria are assessed using MINI interview and Hamilton Depression scale conducted by trained and certified interviewers. Participants may not participate if they are currently completing CBT outside of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2024-09-07 (Actual); Study Completion 2024-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA TMS Clinical and Research Service, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 individuals were recruited and screened
Pre-assignment Details: Excluded (n=60)
  * Not meeting inclusion criteria (n= 9)
  * Declined to participate (n=51)
  * Other reasons (n=0)
  Arm 2 Lost to follow-up (no reason given) (n=4) Discontinued intervention (no reason given (3), COVID diagnosis mid-treatment (1), cited poor fit with intervention (2), repeated non-attendance at scheduled appointments (2), started CBT with outside therapist (1)) (n=9)
Period: Overall Study
Arm/Group | iCBT and TMS | Psychoeducation and TMS
Started | 18 | 18
Completed | 15 | 5
Not Completed | 3 | 13
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iCBT and TMS | Psychoeducation and TMS | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 12 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 17 | 15 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 16 | 14 | 30
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HAM-D)
Description: Change in Depression Symptoms (Range = 0-52, higher indicates greater symptoms)
Time Frame: Baseline to Post-Treatment (6 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCBT and TMS | Psychoeducation and TMS
Number analyzed (Participants) | 18 | 18
score on a scale
  Baseline | 20.4375 (4.0983) | 21.7692 (4.6035)
  6 weeks | 11.3333 (6.6297) | 11.9231 (8.7983)

2. Primary Outcome: Temporal Experience of Pleasure Scale (TEPS)
Description: Change in Depression Symptoms (Range = 0-108, higher indicates lower symptoms)
Time Frame: Baseline to Post-Treatment (6 weeks), as well as 6-month and 9-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCBT and TMS | Psychoeducation and TMS
Number analyzed (Participants) | 18 | 18
score on a scale
  Baseline | 59.1875 (8.8861) | 58.75 (12.9483)
  6 weeks | 61.8125 (12.9523) | 73.5 (9.6658)
  6 months | 65.0833 (13.9705) | 73.3333 (6.6583)
  9 months | 60.8462 (12.8572) | 76 (6.5574)

3. Primary Outcome: Inventory of Depressive Symptomatology (IDS)
Description: Change in Depression Symptoms (Range = 0-78, higher indicates greater symptoms)
Time Frame: Baseline to Post-Treatment (6 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCBT and TMS | Psychoeducation and TMS
Number analyzed (Participants) | 18 | 18
score on a scale
  Baseline | 42.4444 (9.8651) | 42.0556 (12.0317)
  6 weeks | 29.2222 (15.2915) | 25.9412 (14.2279)

4. Primary Outcome: Dimensional Anhedonia Rating Scale (DARS)
Description: Change in Depression Symptoms (Range = 0-130, higher indicates lower symptoms)
Time Frame: Baseline to Post-Treatment (6 weeks), as well as 6-month and 9-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCBT and TMS | Psychoeducation and TMS
Number analyzed (Participants) | 18 | 18
score on a scale
  Baseline | 78.125 (15.5258) | 75 (34.9987)
  6 weeks | 90.2667 (25.401) | 104.1429 (19.4545)
  6 months | 73.3846 (39.7147) | 88.25 (59.1573)
  9 months | 81.0769 (22.4591) | 116.3333 (9.815)

ADVERSE EVENTS:
Time Frame: Adverse events, if had occurred, would be collected during the first 6 weeks of enrollment.
Arm/Group | iCBT and TMS | Psychoeducation and TMS
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT05988619/Prot_SAP_001.pdf